CLINICAL TRIAL: NCT04345250
Title: Bone Response to Exercise Before and After One Week of Energy Restriction in Young Adults
Brief Title: Bone Response to Exercise and Energy Restriction in Young Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was suspended during the COVID-19 pandemic and has not resumed yet.
Sponsor: Brock University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Panagiota Klentrou, Professor, Brock University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 19-247
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Bone Resorption; Bone Loss
Keywords: bone; biomarkers; cycling; diet; youth; females
MeSH Terms: conditions — Bone Resorption; Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Single group, pre to post one week intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): For a period of 6 days between the exercise trials (i.e., following visit 3), each participant will be put on a restricted energy restricted diet consisting of a 25% reduction in their habitual total daily calorie intake. To keep the diet consistent and standardized, participants will record their typical food intake during a control week using the "Eat This Much" app, which will then provide an overall portion plan and the 25% caloric restriction measure for the intervention week. Thus, the intervention diet will mirror the control diet in terms of types of food consumed, with the difference being in the amount consumed. There will be no restriction regarding water, but drinks will be restricted according to the overall calorie intake plan.
  Interventions: Other: Energy restriction

INTERVENTIONS:
Other: Energy restriction — A 25% reduction in total caloric intake, as calculated through the app. Therefore, during the control period, participants will input what they consume into the Eat This Much app, then the app will calculate the 25% reduction in calories to present participants with how much to consume of the same foods. By doing this their diet will not be altered in terms of macronutrients or micronutrients, but solely on calories.

SUMMARY:
Cycling is commonly questioned whether it provides adequate mechanical strain on bone as many elite cyclists have been found to have a low bone mass. However, it remains unclear if this is due to cycling or low energy availability. In addition, acute dietary energy restriction has been found to be accompanied by an imbalance in bone remodelling with reduced bone formation. The objective of this proposal is to examine whether short-term energy restriction leads to changes in markers of bone formation and resorption at rest and in response to cycling in young adults. Specifically, the study will examine changes in circulating bone markers in 15 males and females (ages 18-24) both at rest and following one 45-minute spinning class both before and after one week of restricted energy intake. Blood will be drawn at rest (pre-trial, fasted), and 3 times post-trial (5 min, 1h and 24h); then analysed for biochemical markers of bone formation (BAP and OPG) and resorption (CTX and RANKL) to assess the impact of energy restriction on bone at rest and in response to exercise. This innovative work has potential to make significant advances in understanding tissue growth and development in response to exercise and malnutrition.

DETAILED DESCRIPTION:
Introduction: The skeletal system serves a variety of purposes such as providing structural support, locomotion, protection and more. In order to sustain these functions, bone strength must be upheld. The process of replacing older, microdamaged bone with newer, healthier bone is known as bone remodelling. Bone remodelling involves the balance/coupling of bone resorption and bone formation. Mechanical loading is the magnitude of stress placed on the bone that stimulates bone remodelling, which determines bone mineral density (BMD) and promotes bone growth (Olmedillas et al. 2011). Thus, human research on the determinants of bone growth and strength, is focused on two common factors, exercise and nutrition. Although cycling, a predominantly aerobic exercise, is exceptional for cardiovascular fitness, it is commonly questioned whether it provide adequate mechanical strain on bone. To date the literature surrounding cycling and its impact on bone is contradicting and limited. Inadequate energy intake may also influence BMD via reductions in bone mineral content. Energy restriction is known to reduce insulin-like growth factor 1 (IGF-1), which plays an important role in bone formation 5. Acute dietary energy restriction has been found to be accompanied by an imbalance of bone remodelling with reduced bone formation, which is especially dangerous in aerobic sports that expend a great amount of energy, such as cycling. Many professional and master cyclists are classified as osteopenic (Medelli et al. 2000). Specifically, female cyclists have shown significant lower values of whole-body BMD, and a lower bone strength, than male cyclists (Olmedillas et al. 2011). In addition, female cyclists are known to be energy deficient (low calorie intake) with the average energy intake being 85% of the Recommended Dietary Allowance (RDA). Therefore, it is important to understand whether cycling is a poor form of exercise for bone health or whether the energy restriction, alone or in combination with cycling, is the true underlining issue.

Objective: The objective of this study is to examine whether short-term energy restriction leads to changes in markers of inflammation, oxidative stress, bone turnover at rest and in response to cycling in young adults. Specifically, the study will examine changes in circulating bone markers at rest and following one bout of low impact 45-minute spinning (cycling) both before and after one week of restricted energy intake.

Methods: Fifteen healthy males and females, aged 20-25 years, will be invited to participate in this study, which involves one control trial and two exercise trial visits scheduled one week apart. Females will be on monophasic oral contraceptives, During the control trial, participants will be briefed on the purpose and procedures, will fill out an exercise screening questionnaire, and will provide 4 resting blood samples. One week later, participants will perform the first exercise trial of one 45 minute spin session. Following the first trial, the participants will go on a predetermined energy deficient diet (25% of their habitual diet) for one week, at the end of which they will perform the second trial following the same cycling protocol. Between the first and last visit the participants will be receiving a Fitbit to monitor their activity (steps, heart rate, physical activity participation) and nutritional habits in a food log. To keep the diet consistent and standardized, participants will also be asked to record their habitual food intake during the control week using the "Eat This Much" app, which will provide an overall portion plan and a 25% caloric restriction measure for the intervention week. Thus, the intervention diet will mirror the control diet in terms of types of food consumed, with the difference being in the amount consumed. There will be no restriction regarding water, but drinks will be restricted according to the overall calorie intake plan.In both trials, blood will be drawn at rest (i.e., pre-trial, fasted), and 3 times post-trial (5 min, 1h and 24h). The blood will be centrifuged and the serum separated, aliquoted and then stored at -80 °C until analysis 8. The serum will be analysed for biochemical markers of bone turnover (e.g. osteocalcin, bone-specific alkaline phosphatase [BAP]; osteoprotegerin [OPG]) and bone resorption (C-telopeptides of type I collagen [CTX]; receptor activator of nuclear factor κB ligand [RANKL], sclerostin) to assess the impact of energy restriction on bone at rest and in response to exercise. Metabolic and oxidative stress markers, inflammatory cytokines, adipokines, growth factors and hormones will also be assessed to examine potential mediating effects.

Impact: This innovative work has the potential to make significant advances in understanding the impact of energy restriction and cycling on bone health. The findings from this work will be translatable to understanding tissue growth and development in response exercise and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males and females, aged 20 to 25 years
* healthy (not suffering from asthma)
* without any fracture over the last year
* not taking any medication related to a chronic condition or bone health including food/nutritional supplements (e.g. protein, vitamin D, calcium)
* nonsmokers
* females on monophasic oral contraceptives.

Exclusion Criteria:

* Injuries or chronic conditions in which exercise may pose a risk (e.g., ACL or knee/hip/lower back injuries, arthritis, osteoporosis, neuromuscular diseases)
* any restrictive food allergies or dietary restrictions that would require alterations to the diet plan (i.e, vegan, vegetarian) and or
* any eating disorders (e.g., bulimia, and or anorexia)

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Bone turnover marker | one week
  Osteocalcin in ng/ml
Bone formation marker | one week
  Bone-specific alkaline phosphatase [BAP] in ng/ml
Bone resorption marker | one week
  C-telopeptides of type I collagen [CTX] in ng/ml
Bone formation osteokine | one week
  Osteoprotegerin [OPG] in ng/ml
Bone resorption osteokine | one week
  Receptor activator of nuclear factor κB ligand [RANKL] in ng/ml
Wnt signaling related osteokine | one week
  Sclerostin in ng/ml
Anti-inflammatory cytokine | one week
  Interleukin 10 [IL-10] in pg/ml
Pro-inflammatory cytokine | one week
  Tumor necrosis factor alpha (TNF-α) in pg/ml
Myokine | one week
  Interleukin 6 [IL-6] in pg/ml
Irisin | one week
  Irisin in pg/ml
Oxidative stress marker | one week
  protein carbonyls (PC) in mmol/mg serum protein

SECONDARY OUTCOMES:
Body mass | one week
  Total body mass in kg
Lean body mass | one week
  Fat-free mass in kg
Fat body mass | one week
  Fat mass in kg

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Klentrou, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olmedillas H, Gonzalez-Aguero A, Moreno LA, Casajus JA, Vicente-Rodriguez G. Bone related health status in adolescent cyclists. PLoS One. 2011;6(9):e24841. doi: 10.1371/journal.pone.0024841. Epub 2011 Sep 30. PMID 21980360
- [Background] Medelli J, Lounana J, Menuet JJ, Shabani M, Cordero-MacIntyre Z. Is osteopenia a health risk in professional cyclists? J Clin Densitom. 2009 Jan-Mar;12(1):28-34. doi: 10.1016/j.jocd.2008.07.057. Epub 2008 Oct 1. PMID 18835799